CLINICAL TRIAL: NCT01377792
Title: Phase 4 Study of the Efficacy of Long-term Treatment With Hypertonic Saline on Pulmonary Exacerbations in Patients With Cystic Fibrosis
Brief Title: Study of Long-term Treatment With Hypertonic Saline in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Adelaida Lamas Ferreiro (Other)
Responsible Party: Sponsor-Investigator, Adelaida Lamas Ferreiro, Dra.Adelaida Lamas Ferreiro, Hospital Universitario Ramon y Cajal
Organization: Hospital Universitario Ramon y Cajal (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSH-FQ1
Record Dates: First submitted 2011-05-09; First posted 2011-06-21 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Cystic Fibrosis
Keywords: hypertonic saline; cystic fibrosis; pulmonary inflammation; pulmonary exacerbation
MeSH Terms: conditions — Cystic Fibrosis; Pneumonia | interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5 ml (Active Comparator)
  Interventions: Drug: Hypertonic saline
- 10 ml (Active Comparator)
  Interventions: Drug: Hypertonic saline

INTERVENTIONS:
Drug: Hypertonic saline — comparison of different dosages of drug

SUMMARY:
A phase IV clinical trial, multicentric (3 Hospitals in Madrid) controlled, prospective, open and randomized of long-term treatment with hypertonic saline in cystic fibrosis patients. The purpose of this study is to verify if the long term inhalation (48 weeks) of major volume (10 ml) increases the free time without pulmonary exacerbation, and if this increase is superior to the obtained with the inhalation of the standard volume (5 ml) that has been advocated.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Cystic fibrosis
* Over 6 years old
* FEV1 over than 30%
* Must be able to perform a spirometry
* Must be able to perform induced sputum
* Must tolerate the maximum dose of 10 ml hypertonic saline
* No oral neither intravenous treatment within the previous 2 weeks before the beginning of the study
* No treatment with hypertonic saline in the 2 weeks before

Exclusion Criteria:

* No clinical diagnosis of Cystic Fibrosis
* No tolerance of 10 ml of hypertonic saline
* Positive pregnancy test
* No tolerance of Beta2-agonist
* Treatment with corticosteroids
* FEV1 < 30%
* Liver and/or lung transplantation
* Oxygen treatment
* Hospital admission within the 4 previous weeks
* Oral or intravenous antibiotic treatment within the 2 previous weeks
* Smokers
* Pulmonary colonisation with Burkholderia cepacia complex

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2009-03; Primary Completion 2011-05 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Free time, specified in days, of pulmonary exacerbation | 12 months
  Exact number of days, along 48 weeks of tretment with hypertonic saline, in wich the patient is free of pulmonary excaerbation symptoms and does not need antibiotics.

SECONDARY OUTCOMES:
Changes in lung function test measured by spirometry | 12 months
Changes in inflammatory markers during the treatment | 12 months
  Measurement of inflammatory markers in induced sputum.
Quality of life | 12 months
  Measurement of quality of life of patients during treatment by CFQ-R test

CONTACTS AND LOCATIONS:
Overall Officials: Adelaida Lamas, MD, Principal Investigator
Locations (1):
- Cystic Fibrosis Unit. Ramón y Cajal University Hospital, Madrid, Madrid, Spain